CLINICAL TRIAL: NCT07383701
Title: Lactiplantibacillus Plantarum 299v Probiotic Probiotic Supplementation in Patients With Diabetic Macular Edema
Brief Title: Lactiplantibacillus Plantarum 299v Probiotic Supplementation in Patients With Diabetic Macular Edema
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Demetrios Vavvas, Solman and Libe Friedman Professor of Ophthalmology Director Retina Service Mass. Eye and Ear / Mass General Hospital Co-Director Ocular Regenerative Medical Institute Harvard Medical School, Massachusetts Eye and Ear Infirmary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025P001157
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Macular Edema
Keywords: diabetic macular edema; Lactiplantibacillus plantarum 299v; probiotic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Main Arm - twice daily for 4 months (Experimental): This is the only arm in this study. All participants will receive 4 months of Lactobacillus plantarum supplementation.
  Interventions: Drug: Lactobacillus plantarum 299v

INTERVENTIONS:
Drug: Lactobacillus plantarum 299v — Lactiplantibacillus Plantarum 299v Probiotic Supplementation, Twice Daily, for 4 Months

SUMMARY:
In this pilot prospective, interventional, longitudinal study, we aim to evaluate the potential benefits of the probiotic supplement Lactobacillus plantarum 299v in patients with diabetic macular edema (DME).

The study seeks to address the following questions:

1. Does central macular thickness on optical coherence tomography decrease after 4 months of supplementation?
2. Is visual acuity improved at 1, 2, 3, and 4 months following initiation of supplementation?
3. Is the number of anti-VEGF injections reduced following initiation of supplementation?

Outcomes will be compared to a control group, using historic retrospective data.

Participants will take Lactobacillus plantarum 299v orally twice daily for four months.

DETAILED DESCRIPTION:
Study Design: Prospective open label longitudinal interventional study with oral probiotic supplement Lactobacillus plantarum.

Inclusion criteria: Age of at least 18 years, presence of DME at the current clinical visit

Exclusion criteria: Patients with contraindication to probiotic supplement (e.g. prior allergy or GI intolerance and any type of immunocompromised diseases).

Eligible individuals (patients at least 18 years old with diabetic macular

Participants: Patients with DME that belong in the following two groups:

* Group A: 12 Patients with mild DME and good visual acuity (<= 20/30) similar to DRCR network protocol V that do not need anti-VEGF injections as per standard clinical care.
* Group B: 12 Patients with DME that need anti-VEGF injections as per standard clinical care.

Intervention: Oral probiotic supplement L. plantarum 299v twice daily for 4 months for both groups.

Study outcomes:

* OCT with central macular thickness (CMT) at 1, 2, 3, 4-months follow-up.
* Visual Acuity at 1, 2, 3, 4-months follow-up.
* Number of anti VEGF injections.

In group A, we aim to measure what percentage of patients with a stability or improvement in DME as determined by a stability (+/- 9% of OCT CMT) or a reduction of DME (>= 30 microns or >= 10% decrease of CMT) from baseline. Secondary endpoints will be visual acuity and need for injection initiation during the 4 months.

In group B we will measure same outcomes as in group A. Furthermore, we aim to measure the number of injections that these DME patients will need over the course of 4 months.

For both groups we will also investigate whether the addition of the probiotic supplement altered the course of disease compared to historical data.

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 18 years, presence of DME at the current clinical visit

Exclusion Criteria:

* Patients with contraindication to probiotic supplement (e.g. prior allergy or GI intolerance and any type of immunocompromised diseases).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Central Macular Thickness | 1,2,3,4-months following supplement initiation
  Central macular thickness (CMT) on optical coherence tomography

SECONDARY OUTCOMES:
Best corrected visual acuity | 1, 2, 3, 4-months following supplement initiation
  Best corrected visual acuity
Anti-VEGF Frequency | At 1,2,3,4-months following supplement initiation
  Number of anti VEGF injections

CONTACTS AND LOCATIONS:
Locations (1):
- Mass Eye and Ear, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Although data would be de-identified, the small sample size and single-center design increase the risk of re-identification. Therefore, results will be reported in aggregate only. There are no current plans for external sharing of IPD.

REFERENCES:
- [Result] Senger DR, Li D, Jaminet SC, Cao S. Activation of the Nrf2 Cell Defense Pathway by Ancient Foods: Disease Prevention by Important Molecules and Microbes Lost from the Modern Western Diet. PLoS One. 2016 Feb 17;11(2):e0148042. doi: 10.1371/journal.pone.0148042. eCollection 2016. PMID 26885667
- [Result] Kensler TW, Wakabayashi N, Biswal S. Cell survival responses to environmental stresses via the Keap1-Nrf2-ARE pathway. Annu Rev Pharmacol Toxicol. 2007;47:89-116. doi: 10.1146/annurev.pharmtox.46.120604.141046. PMID 16968214
- [Result] Li JQ, Welchowski T, Schmid M, Letow J, Wolpers C, Pascual-Camps I, Holz FG, Finger RP. Prevalence, incidence and future projection of diabetic eye disease in Europe: a systematic review and meta-analysis. Eur J Epidemiol. 2020 Jan;35(1):11-23. doi: 10.1007/s10654-019-00560-z. Epub 2019 Sep 12. PMID 31515657